CLINICAL TRIAL: NCT02483949
Title: Healthy Eating and Active Living for Diabetes - Gestational Diabetes Mellitus
Acronym: HEALD-GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athabasca University (Other)
Responsible Party: Principal Investigator, Steven T. Johnson, Assistant Professor, Athabasca University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEALD-GDM
Record Dates: First submitted 2015-05-28; First posted 2015-06-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Gestational Previous Pregnancy
MeSH Terms: interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): Lifestyle intervention with peer-counseling follow-up
  Interventions: Behavioral: Healthy Eating and Active Living for Diabetes - Gestational Diabetes Mellitus

INTERVENTIONS:
Behavioral: Healthy Eating and Active Living for Diabetes - Gestational Diabetes Mellitus
  Other Names: HEALD-GDM
  Arms: Intervention

SUMMARY:
To examine the effectiveness of a group-based lifestyle modification program followed by peer-led telephone counselling for type 2 diabetes (T2D) and cardiovascular disease risk reduction. The lifestyle modification program will support daily ambulatory activity and low glycemic index food intake among women with previous gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Study Objective:

To examine the effectiveness of a group-based lifestyle modification program followed by peer-led telephone counselling for type 2 diabetes (T2D) and cardiovascular disease risk reduction. The lifestyle modification program will support daily ambulatory activity and low glycemic index food intake among women with previous GDM.

Methods:

To achieve the study objective, the HEALD-GDM lifestyle modification program already proven effective for adults with T2D among women with previous GDM within 12 months postpartum will be evaluated. Women will take part in either the HEALD-GDM program (intervention) or in usual care (control). To evaluate the effectiveness of HEALD-GDM, a randomized, two-arm, before and after study design is proposed. Potentially eligible participants will be recruited from Diabetes in Pregnancy Clinics in Calgary and Edmonton, Alberta. Following identification of eligible participants, the investigators will randomize 100 participants to either the HEALD-GDM program or to usual care control (i.e., 50 per group). A Canadian Society of Exercise Physiology certified instructor (Exercise Specialist) trained in HEALD-GDM delivery will lead the program. Group-based classes will be held at community recreational centres in Calgary and Edmonton (one site each) in months one and four of the 24-week HEALD-GDM program. Theory-guided peer-led telephone counselling will supplement the program. HEALD-GDM focuses broadly on T2D prevention through lifestyle modification and will be based on a proven effective pedometer-based active living behaviour.

The primary outcome will be change in objectively measured moderate and vigorous physical activity at assessment appointments (baseline and 24 weeks). Secondary outcomes include: 1) body mass, 2) glycemic control (hemoglobin A1c), 3) musculoskeletal and cardiorespiratory fitness, 4) dietary intake, 5) metabolic biomarkers, 6) health-related quality of life (HRQL), social-cognitive mediators and 7) mental health.

Significance:

Evidence for appropriate lifestyle modification programs for this high-risk population is lacking. This study will serve to inform best practices for diabetes and cardiovascular disease risk reduction through known modifiable risk reduction targets such as healthy eating and active living.

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed previous and recent (within last 12 months) gestational diabetes mellitus • informed consent

Exclusion Criteria:

* unable to provide informed consent or unwilling to participate in the study
* unable to read, understand and converse in English
* contraindications based on the Canadian Society for Exercise Physiology Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* currently enrolled in other diabetes-related research studies
* pregnant or planning another pregnancy in the next 12 months (any participants becoming pregnant at any point during the study will only contribute data prior to their pregnancy date)
* hemoglobin A1c >6.5% or clinical suspicion of type 1 or type 2 diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months of moderate and vigorous physical activity (walking). | 6 months
  Accelerometer derived MVPA

SECONDARY OUTCOMES:
Change from baseline to 6 months in Low Glycemic Index foods. | 6 months
  Low glycemic index food intake will be assessed using three-day food records.

CONTACTS AND LOCATIONS:
Overall Officials: Steven T. Johnson, PhD, Principal Investigator — Athabasca University
Locations (2):
- Canada (2):
  - Athabasca University, Athabasca, Alberta
  - Alliance for Canadian Health Outcomes Research in Diabetes, Edmonton, Alberta

REFERENCES:
- [Derived] Johnson ST, Mladenovic AB, Mathe N, Davenport MH, Butalia S, Qiu W, Johnson JA. Healthy eating and active living after gestational diabetes mellitus (HEALD-GDM): Rationale, design, and proposed evaluation of a randomized controlled trial. Contemp Clin Trials. 2017 Oct;61:23-28. doi: 10.1016/j.cct.2017.07.008. Epub 2017 Jul 9. PMID 28700892
- See also: Funding agency — http://lawson.ca/diabetes